CLINICAL TRIAL: NCT06059001
Title: A Phase 1b Study to Evaluate the Safety, Pharmacokinetics, and Anti-Tumour Activity of the Myc Inhibitor OMO-103 Administered Intravenously in Patients With Advanced Solid Tumours
Brief Title: Study to Evaluate the Safety, PK, and Efficacy of the Myc Inhibitor OMO-103 Administered iv in Patients With PDAC
Acronym: OMO-103-02
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peptomyc S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMO-103-02
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: PDAC; Pancreatic cancer; metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-Paclitaxel+Gemcitabine+OMO-103 (Experimental): SoC Gemcitabine/Nab-Paclitaxel plus experimental OMO-103
  Interventions: Drug: OMO-103; Drug: Nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: OMO-103 — Investigational Product: 35 mg/mL (4.5 mL/vial) concentrate for solution for infusion
Drug: Nab-Paclitaxel — IV infusion - Standard of Care
Drug: Gemcitabine — IV infusion - Standard of Care

SUMMARY:
This study is an open-label, multicentre, Phase 1b trial designed to determine the safety, tolerability, efficacy, PK, pharmacodynamics (PD) and proof-of-concept of OMO-103 in combination with the standard regimen gemcitabine/nab-paclitaxel in patients with metastatic pancreatic cancer who are treatment-naïve in the advanced disease setting.

DETAILED DESCRIPTION:
This study is an open-label, multicentre, Phase 1b trial designed to determine the safety, tolerability, efficacy, PK, pharmacodynamics (PD) and proof-of-concept of OMO-103 in combination with the standard regimen gemcitabine/nab-paclitaxel in patients with metastatic pancreatic cancer who are treatment-naïve in the advanced disease setting. The study consists of two parts:

Part 1 (Safety-Run-In) in patients with metastatic pancreatic cancer, evaluating OMO-103 plus gemcitabine/nab-paclitaxel in two dose levels at 75% and 100% of the RP2D.

Approximately six patients will be enrolled in Part 1, covering two dose levels with the primary objective of determining the safety and tolerability of OMO-103 plus gemcitabine/nab-paclitaxel and defining an appropriate dose for further evaluation in Part 2.

Part 2 (Dose expansion) in patients with metastatic pancreatic cancer where gemcitabine/nab-paclitaxel is a suitable treatment option. Patients will be treated with the dose found in part 1 to further characterise the safety, tolerability, PK, PD and anti-tumour activity of this combination

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients, 18 years of age or older who sign the ICF and are willing and able to comply with the study protocol.

  2. Histologically or cytologically proven pancreatic cancer (pancreatic ductal adenocarcinoma [PDAC]).

  3. Patients have to be treatment naïve in the metastatic setting (neo-or adjuvant treatment has to be finished at least six months before) and are suitable to receive the standard regimen gemcitabine and nab-paclitaxel.

  4. Patients must show a specific biomarker signature, which will be analysed before inclusion into the study, comprising CD62E, MIP-1ß, MCP-1 and IL-8.

  5. Patients must have measurable disease as per RECIST v1.1 criteria and documented by computed tomography (CT) and/or magnetic resonance imaging (MRI). NOTE: Lesions to be used as measurable disease for the purpose of response assessment must either:
  1. not reside in a field that has been subjected to prior radiotherapy, or
  2. have demonstrated clear evidence of radiographic progression since the completion of prior radiotherapy and prior to study enrolment.

     6. Tumour biopsy (either from the primary tumour or from metastases) during Screening and during Treatment should be obtained from the patients. NOTE: In case a patient has had a tumour biopsy in the previous 6 months and a paraffin block is available, a new biopsy does not need to be done at Screening.

     7. For each patient undergoing pre- and on-treatment biopsies, the identified lesion to be biopsied should not have been previously irradiated and should not be the only lesion being utilised as a measurable-disease target lesion for objective response assessment. Patients must have tumour lesions that can be accessed for biopsy with acceptable clinical risk in the judgement of the Investigator.

     8. ECOG performance status up to 1. 9. Adequate organ function as defined by the following criteria:

     Haematological:

     o Neutrophils ≥1,500/μL

     o Platelets ≥100,000/μL
     * Haemoglobin ≥10 g/dL

     Renal:

     o Creatinine Clearance (calculated via Cockcroft-Gault Equation) ≥50 mL/min

     Hepatic:

     o Serum total bilirubin ≤1.5 upper limit of normal (ULN) or

     o Direct bilirubin ≤ULN for patients with total bilirubin >1.5 ULN

     o Aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic-pyruvic transaminase (ALT/SGPT) ≤2.5 ULN or ≤5 ULN if liver metastases

     Chemistry:
     * Albumin >30 g/L. 10. If not postmenopausal or surgically sterile, female patients must be willing to practice at least one of the following highly effective methods of birth control (defined as having a low failure rate) for at least a menstrual cycle before and for 1 month after last study drug administration:

  <!-- -->

  1. True abstinence, when this is in line with the preferred and usual lifestyle of the patient, from sexual intercourse with a member of the opposite sex;
  2. Sexual intercourse with vasectomised male;
  3. Hormonal female contraceptive (oral, parenteral, intravaginal, implantable or transdermal) for at least 3 consecutive months prior to investigational product administration (when not clinically contraindicated as in breast, ovarian and endometrial cancers);
  4. Use of an intrauterine contraceptive device. 11. Male patients and their sexual partners must use an appropriate contraceptive from Screening for 6 months after last study drug administration, including:

  <!-- -->

  1. True abstinence
  2. Male sterilisation
  3. Hormonal female contraceptive (oral, parenteral, intravaginal, implantable or transdermal) and condom
  4. Intrauterine contraceptive device and condom.

Exclusion Criteria:

1. Systemic anti-cancer therapy within four weeks prior to study drug administration.
2. Radiation therapy within four weeks prior to study entry. Localised palliative radiotherapy to non-target lesions is allowed.
3. Previous or concurrent malignancy that could affect compliance with the protocol or interpretation of results. Patients curatively treated more than 2 years prior to enrolment, and patients with adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ are eligible.
4. Previous treatment with either gemcitabine or nab-paclitaxel in any setting.
5. Contraindication to receive gemcitabine/nab-paclitaxel.
6. Non-malignant systemic disease including cerebrovascular accident, unstable angina pectoris, unstable atrial fibrillation, unstable cardiac arrhythmia, myocardial infarction in the last six months, New York Heart Association (NYHA) Class III or IV heart failure.
7. Patients with active uncontrolled infection or known to be serologically positive for human immunodeficiency virus (HIV), hepatitis B (except after vaccination) or hepatitis C infection. Investigators may test as per their discretion.
8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
9. Pregnant or nursing.
10. Patients with symptomatic or unstable central nervous system primary tumour or metastases and/or carcinomatous meningitis.
11. Live vaccine in the last four weeks.
12. Current participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of AEs, SAEs to evaluate the safety and tolerability of OMO-103 plus gemcitabine/nab-paclitaxel | through study completion, an average of 2 years
  To evaluate the safety and tolerability of OMO-103 plus gemcitabine/nab-paclitaxel in adult patients with metastatic pancreatic cancer being treatment naïve.

SECONDARY OUTCOMES:
To assess the anti-tumour activity of OMO-103 plus gemcitabine/nab-paclitaxel as measured by objective response rate (ORR) | through study completion, an average of 2 years
  ORR, PFS, DCR, TTP, TTR, and DOR assessed via RECIST v1.1 criteria.
Ratio of patients with positive cytokine predictive signature result and its impact on efficacy | through study completion, an average of 2 years
  Predictive cytokine signature and its impact on efficacy (as above)
To assess the anti-tumour activity via 3D-volumetric measurement | through study completion, an average of 2 years
  Percentage of tumour burden change evaluated via 3D volumetric analysis of the total tumour burden.
Type, incidence, severity, timing, seriousness, and relatedness of AEs and laboratory | through study completion, an average of 2 years
  Type, incidence, severity, timing, seriousness, and relatedness of AEs and laboratory abnormalities.
To characterise the PK of OMO-103 plus gemcitabine/nab-paclitaxel | through study completion, an average of 2 years
  PK parameters of OMO-103 plus gemcitabine/nab-paclitaxel
To assess the development of human ADAs to OMO-103. | through study completion, an average of 2 years
  Incidence of ADAs to OMO-103
To evaluate quality of life (QoL) in patients with metastatic pancreatic cancer | through study completion, an average of 2 years
  Scores on the validated European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) (version 3) and QLQ-PAN26 (EORTC PAN26)
  QLQ-PAN26: Scale with values from 1 to 4, where 4 is the most positive for the patient's quality of life.
  QLQ-C30: Scale with values from 1 to 4, where 1 is the most positive for the patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Macarulla, MD, PhD, Principal Investigator — Hospital Vall d´Hebrón
Locations (6):
- Spain (6):
  - Hospital Vall d´Hebrón, Barcelona, Barcelona
  - ICO Hopsitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Regional Universitario de Málaga, Málaga, Spain
  - Hospital Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No